CLINICAL TRIAL: NCT00299546
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Trial of Golimumab, a Fully Human Anti-TNFa Monoclonal Antibody, Administered Subcutaneously in Subjects With Active Rheumatoid Arthritis and Previously Treated With Biologic Anti- TNFa Agent(s)
Brief Title: A Study of the Safety and Efficacy of Golimumab (CNTO 148) in Subjects With Active Rheumatoid Arthritis Previously Treated With Biologic Anti-TNFa Agent(s)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR006334; C0524T11 (Other: Centocor)
Record Dates: First submitted 2006-03-03; First posted 2006-03-07 (Estimated); Results first posted 2011-09-28 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-01

CONDITIONS: Arthritis, Rheumatoid
Keywords: Rheumatoid Arthritis; Anti-TNFa agents; subcutaneous injection
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — golimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1: Placebo (Placebo Comparator): Placebo Subcutaneous (SC) injections every 4 weeks (wks) thru Wk 20 (unless early escape at Wk 16); Golimumab - if early escape, 50 mg SC injections from Wk 16 up to 5 yrs; Golimumab - 50 mg SC injections beginning Wk 24 up to 5 yrs (unless early escape); Golimumab - Dr's discretion after unblinding, dose adjusted from 50 to 100 mg and from 100 to 50mg. Duration of the blinded period will be until the week-24 database lock.
  Interventions: Drug: Placebo; Biological: Golimumab 50 mg
- Group 2: Golimumab 50 mg (Experimental): Golimumab 50 mg SC injections every 4 wks from Wk 0 up to 5 yrs (unless early escape at Wk 16); Golimumab - if early escape, 100 mg SC injections every 4 wks beginning Wk 16 up to 5 yrs; Golimumab - Dr's discretion after unblinding, dose adjusted from 50 to 100 mg and from 100 to 50mg. Duration of the blinded period will be until the week-24 database lock.
  Interventions: Biological: Golimumab 50 mg
- Group 3: Golimumab 100 mg (Experimental): Golimumab 100 mg SC injections every 4 wks from Wk 0 up to 5 yrs; Golimumab - Dr's discretion after unblinding, dose adjusted from 100 to 50 mg. Duration of the blinded period will be until the week-24 database lock.
  Interventions: Biological: Golimumab 100 mg

INTERVENTIONS:
Drug: Placebo — SC injections
  Arms: Group 1: Placebo
Biological: Golimumab 50 mg — SC injections
  Arms: Group 1: Placebo; Group 2: Golimumab 50 mg
Biological: Golimumab 100 mg — SC injections
  Arms: Group 3: Golimumab 100 mg

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of golimumab (CNTO 148) in subjects who have active rheumatoid arthritis and have been treated previously with at least 1 dose of a biologic anti-TNFa agent (etanercept, adalimumab or infliximab).

DETAILED DESCRIPTION:
Golimumab is a fully human protein (antibody) which binds to tumor necrosis factor-alpha (TNFa). TNFa is increased in patients with rheumatoid arthritis (RA), and plays a major role in causing the joint pain, swelling and damage from RA. Other marketed drugs that target TNFa (anti-TNFa drugs) have been shown to be effective in reducing the symptoms, signs and joint damage of RA, but have limitations with respect to safety and ease of use. This is a randomized, double-blind, placebo-controlled trial of the efficacy and safety of a new anti-TNFa drug, golimumab, at 2 doses, injected under the skin every 4 weeks in subjects with active RA previously treated with at least 1 dose of a biologic anti-TNFa agent (etanercept, adalimumab or infliximab). Concomitant therapy with methotrexate, sulfasalazine and/or hydroxychloroquine is permitted if the subject has tolerated these medications for at least 12 weeks prior to the first administration of study drug and is on a stable dose for at least 4 weeks prior to the first administration of study agent. The study hypothesis is that golimumab will be a safe and effective treatment for RA in subjects with active RA previously treated with at least one biologic anti-TNFa agent as measured by the American College of Rheumatology (ACR) response criteria, the Disease Activity Score 28 (DAS28) responses and the change from baseline in Health Assessment Questionnaire (HAQ), without causing unacceptable significant adverse effects. The ACR response criteria were designed to assess the level of improvement in the signs and symptoms of RA. The DAS28 responses also measure improvement in the signs and symptoms of RA using the joint examination and laboratory testing. The HAQ is a series of questions that measure a subject's impairment in physical function caused by RA. Patients will receive golimumab 50 mg or 100 mg or placebo injections under the skin every 4 weeks until Week 24. After Week 24, all subjects receive golimumab 50 mg or 100 mg injections, and golimumab continues for all groups every 4 weeks for about 4 and a half more years.

ELIGIBILITY:
Inclusion Criteria:

* Patients have a diagnosis of rheumatoid arthritis (RA) (according to the revised 1987 criteria of the ACR) for at least 3 months prior to screening
* Have active RA as defined by persistent disease activity with at least 4 swollen and 4 tender joints, at the time of screening and baseline
* Must have been previously treated with at least one dose of etanercept, adalimumab, or infliximab
* If currently using methotrexate, sulfasalazine and/or hydroxychloroquine must have tolerated these agents for at least 12 weeks and be on a stable dose for at least 4 weeks prior to the first administration of study agent
* If using NSAIDs or other analgesics must be on a stable dose for at least 2 weeks prior to the first administration of study agent
* If using oral corticosteroids must be on a stable dose equivalent to <= 10 mg of prednisone/day for at least 2 weeks prior to first administration of study agent
* Are considered eligible according to specified tuberculosis (TB) screening criteria.

Exclusion Criteria:

* Patients cannot have other inflammatory diseases other than RA that might interfere with the evaluation of the benefit of golimumab therapy
* No history of treatment with natalizumab, rituximab or cytotoxic agents
* No history of demyelinating diseases such as multiple sclerosis or optic neuritis or of concurrent congestive heart failure (CHF), lymphoproliferative disease, known malignancy or history of malignancy within the previous 5 years (with the exception of a nonmelanoma skin cancer that has been treated with no evidence of recurrence)
* No history of, or ongoing, chronic or recurrent infectious disease
* No serious infection within 2 months prior to first administration of study agent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 461 (Actual)
Dates: Start 2006-02; Primary Completion 2007-08 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.
Locations (77):
- United States (40):
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Paradise Valley, Arizona
  - La Jolla, California
  - Los Angeles, California
  - Santa Monica, California
  - Torrance, California
  - Upland, California
  - Trumbull, Connecticut
  - Aventura, Florida
  - Jacksonville, Florida
  - Jupiter, Florida
  - Largo, Florida
  - Palm Harbor, Florida
  - Tamarac, Florida
  - Moline, Illinois
  - Springfield, Illinois
  - Cedar Rapids, Iowa
  - Witchita, Kansas
  - Louisville, Kentucky
  - Wheaton, Maryland
  - Boston, Massachusetts
  - Rochester, Minnesota
  - St Louis, Missouri
  - Syracuse, New York
  - Charlotte, North Carolina
  - Wilmington, North Carolina
  - Cincinnati, Ohio
  - Mayfield, Ohio
  - Duncansville, Pennsylvania
  - Pittsburgh, Pennsylvania
  - West Reading, Pennsylvania
  - Knoxville, Tennessee
  - Fort Worth, Texas
  - Houston, Texas
  - Lubbock, Texas
  - Arlington, Virginia
  - Spokane, Washington
  - Brookfield, Wisconsin
  - Racine, Wisconsin
- Australia (3):
  - Adelaide
  - Cotton Tree
  - Melbourne
- Austria (3):
  - Graz
  - Lainz/Wien N/A
  - Vienna
- Canada (9):
  - Victoria, British Columbia
  - Winnipeg, Manitoba
  - St. John's, Newfoundland and Labrador
  - Kitchener, Ontario
  - Newmarket, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Sainte-Foy, Quebec
  - Claire
- Finland (3):
  - Helsinki
  - Hyvinkää
  - Jyvalskyla
- Germany (9):
  - Baden-Baden
  - Berlin
  - Cologne
  - Erlangen
  - Hamburg
  - Herne
  - München
  - Vogelsang-Gommern
  - Würzburg
- Maastricht, Netherlands
- New Zealand (3):
  - Auckland
  - Rotorua
  - Timaru
- Spain (3):
  - Santander
  - Seville
  - Valencia
- United Kingdom (3):
  - Leeds
  - London
  - Oxford

REFERENCES:
- [Derived] Vieira MC, Zwillich SH, Jansen JP, Smiechowski B, Spurden D, Wallenstein GV. Tofacitinib Versus Biologic Treatments in Patients With Active Rheumatoid Arthritis Who Have Had an Inadequate Response to Tumor Necrosis Factor Inhibitors: Results From a Network Meta-analysis. Clin Ther. 2016 Dec;38(12):2628-2641.e5. doi: 10.1016/j.clinthera.2016.11.004. Epub 2016 Nov 24. PMID 27889300
- [Derived] Kay J, Fleischmann R, Keystone E, Hsia EC, Hsu B, Zhou Y, Goldstein N, Braun J. Five-year Safety Data from 5 Clinical Trials of Subcutaneous Golimumab in Patients with Rheumatoid Arthritis, Psoriatic Arthritis, and Ankylosing Spondylitis. J Rheumatol. 2016 Dec;43(12):2120-2130. doi: 10.3899/jrheum.160420. Epub 2016 Nov 1. PMID 27803138
- [Derived] Smolen JS, Kay J, Doyle M, Landewe R, Matteson EL, Gaylis N, Wollenhaupt J, Murphy FT, Xu S, Zhou Y, Hsia EC. Golimumab in patients with active rheumatoid arthritis after treatment with tumor necrosis factor alpha inhibitors: findings with up to five years of treatment in the multicenter, randomized, double-blind, placebo-controlled, phase 3 GO-AFTER study. Arthritis Res Ther. 2015 Jan 22;17(1):14. doi: 10.1186/s13075-015-0516-6. PMID 25627338
- [Derived] Smolen JS, Kay J, Doyle MK, Landewe R, Matteson EL, Wollenhaupt J, Gaylis N, Murphy FT, Neal JS, Zhou Y, Visvanathan S, Hsia EC, Rahman MU; GO-AFTER study investigators. Golimumab in patients with active rheumatoid arthritis after treatment with tumour necrosis factor alpha inhibitors (GO-AFTER study): a multicentre, randomised, double-blind, placebo-controlled, phase III trial. Lancet. 2009 Jul 18;374(9685):210-21. doi: 10.1016/S0140-6736(09)60506-7. Epub 2009 Jun 26. PMID 19560810

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 461 participants were enrolled at 86 sites in North America, Europe, Australia and New Zealand.
Groups:
- Group 1: Placebo: Placebo Subcutaneous (SC) injections every 4 weeks (wks) thru Wk 20 (unless early escape at Wk 16); Golimumab - if early escape, 50 mg SC injections from Wk 16 up to 5 yrs; Golimumab - 50 mg SC injections beginning Wk 24 up to 5 yrs (unless early escape); Golimumab - Dr's discretion after unblinding, dose adjusted from 50 to 100 mg and from 100 to 50mg. Duration of the blinded period was until the week-24 database lock.
- Group 2: Golimumab 50 mg: Golimumab 50 mg SC injections every 4 wks from Wk 0 up to 5 yrs (unless early escape at Wk 16); Golimumab - if early escape, 100 mg SC injections every 4 wks beginning Wk 16 up to 5 yrs; Golimumab - Dr's discretion after unblinding, dose adjusted from 50 to 100 mg and from 100 to 50mg. Duration of the blinded period was until the week-24 database lock.
- Group 3: Golimumab 100 mg: Golimumab 100 mg SC injections every 4 wks from Wk 0 up to 5 yrs; Golimumab - Dr's discretion after unblinding, dose adjusted from 100 to 50 mg. Duration of the blinded period was until the week-24 database lock.
Period: Overall Study
Arm/Group | Group 1: Placebo | Group 2: Golimumab 50 mg | Group 3: Golimumab 100 mg
Started | 155 | 153 | 153
Completed | 55 | 61 | 67
Not Completed | 100 | 92 | 86
Not completed — Death | 3 | 2 | 0
Not completed — Lost to Follow-up | 2 | 2 | 5
Not completed — Adverse Event | 37 | 22 | 27
Not completed — Unsatisfactory therapeutic effect | 34 | 39 | 34
Not completed — Other | 24 | 26 | 19
Not completed — Not treated | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Placebo | Group 2: Golimumab 50 mg | Group 3: Golimumab 100 mg | Total
Number analyzed (Participants) | 155 | 153 | 153 | 461
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (13.07) | 53.9 (11.47) | 53.7 (12.26) | 54.1 (12.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 132 | 113 | 122 | 367
  Male | 23 | 40 | 31 | 94

OUTCOME MEASURES:

1. Primary Outcome: American College of Rheumatology (ACR) 20 Response at Week 14.
Description: ACR 20 response is an improvement of >= 20% from baseline in both the tender and swollen joint count and in at least 3 of the 5 assessments ( patient's assessment of pain visual analog scale (VAS), patient's global assessment of disease activity VAS scale, Physician's global assessment of disease activity VAS scale, Health Assessment Questionnaire and C-reactive protein)
Time Frame: Week 14
Population: Randomized participants (excluding 1 site). Participants considered non-responders if used any prohibited medications or discontinued subcutaneous study agent due to lack of efficacy. Missing ACR components imputed by Last Observation Carried Forward unless all ACR components were missing; in which case considered non-responders.
Measure: Number; unit: participants
Groups:
- Group 1: Placebo: Placebo Subcutaneous (SC) injections every 4 weeks (wks) thru Wk 20 (unless early escape at Wk 16); golimumab - if early escape, 50 mg SC injections from Wk 16 up to 5 yrs; golimumab - 50 mg SC injections beginning Wk 24 up to 5 yrs (unless early escape); golimumab - Dr's discretion after unblinding, dose adjusted from 50 to 100 mg. Duration of the blinded period was until the week-24 database lock.
- Group 2: Golimumab 50 mg: Golimumab 50 mg SC injections every 4 wks from Wk 0 up to 5 yrs (unless early escape at Wk 16); golimumab - if early escape, 100 mg SC injections every 4 wks beginning Wk 16 up to 5 yrs; golimumab - Dr's discretion after unblinding, dose adjusted from 50 to 100 mg. Duration of the blinded period was until the week-24 database lock.
- Combined Golimumab: Combines Group 2 (golimumab 50 mg) and Group 3 (golimumab 100 mg).
Arm/Group | Group 1: Placebo | Group 2: Golimumab 50 mg | Group 3: Golimumab 100 mg | Combined Golimumab
Number analyzed (Participants) | 150 | 147 | 148 | 295
participants | 27 | 51 | 54 | 105
Statistical Analysis 1: Comparison: Group 1: Placebo vs Combined Golimumab; Null hypothesis: No difference in ACR 20 response at Wk 14 comparing Group 1 vs. Combined Groups 2 and 3. A sample size of 140 patients per group provides a >90% power assuming 50% of patients used Methotrexate (MTX) at baseline and 30% ACR 20 response in placebo and 40~55% ACR 20 response in golimumab groups; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — A positive test is concluded if there is a significant difference between combined golimumab and placebo groups and at least one of the pair-wise comparisons at 0.05 level; Stratified by baseline Methotrexate (MTX)
Statistical Analysis 2: Comparison: Group 1: Placebo vs Group 2: Golimumab 50 mg; Null Hypothesis: No difference in ACR 20 response at Wk 14 between Group 1: Placebo and Group 2: 50 mg; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel — Test was performed because Group 1: Placebo was significantly different from Combined Groups 2 & 3; Stratified by baseline MTX
Statistical Analysis 3: Comparison: Group 1: Placebo vs Group 3: Golimumab 100 mg; Null Hypothesis: No difference in ACR 20 response at Wk 14 between Group 1: Placebo and Group 3 :100 mg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Test was performed because Group 1: Placebo was significantly different from Combined Groups 2 & 3; Stratified by baseline MTX

2. Secondary Outcome: American College of Rheumatology (ACR) 50 Response at Week 14
Description: Number of patients who achieved an ACR 50 response at Week (Wk) 14. ACR 50 response is an improvement of >= 50% from baseline in both the tender and swollen joint count and in at least 3 of the 5 assessments ( patient's assessment of pain visual analog scale (VAS), patient's global assessemnt of disease activity VAS scale, Physician's global assessment of disease activity VAS scale, Health Assessment Questionnaire and C-reactive protein).
Time Frame: Week 14
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Group 1: Placebo | Group 2: Golimumab 50 mg | Group 3: Golimumab 100 mg | Combined Golimumab
Number analyzed (Participants) | 150 | 147 | 148 | 295
participants | 10 | 22 | 27 | 49
Statistical Analysis 1: Comparison: Group 1: Placebo vs Combined Golimumab; Test type: Superiority or Other; p = 0.003, Cochran-Mantel-Haenszel; Stratified by baseline Methotrexate (MTX)
Statistical Analysis 2: Comparison: Group 1: Placebo vs Group 2: Golimumab 50 mg; Test type: Superiority or Other; p = 0.021, Cochran-Mantel-Haenszel — Test was performed because Group 1: Placebo was significantly different from Combined Groups 2 & 3; Stratified by baseline MTX
Statistical Analysis 3: Comparison: Group 1: Placebo vs Group 3: Golimumab 100 mg; Test type: Superiority or Other; p = 0.002, Cochran-Mantel-Haenszel — Test was performed because Group 1: Placebo was significantly different from Combined Groups 2 & 3; Stratified by baseline MTX

3. Secondary Outcome: Disease Activity Index Score 28 (DAS 28) (Using C-reactive Protein) Response at Week 14
Description: DAS 28 using C-reactive protein (CRP) is an index to measure disease activity in participants with rheumatoid arthritis which combines tender joint count (28 joints), swollen joint count (28 joints), CRP value, and participant's global assessment of disease activity (using a Visual Analog Scale of 0 to 100 mm). The DAS 28 score ranges from 0 (best) to 10 (worst).
Time Frame: Week 14
Population: Randomized participants (excluding 1 site). Participants considered non-responders if used any prohibited medications or discontinued subcutaneous study agent due to lack of efficacy. Missing DAS 28 components imputed by Last Observation Carried Forward unless all components were missing; in which case considered non-responders.
Measure: Number; unit: participants
Arm/Group | Group 1: Placebo | Group 2: Golimumab 50 mg | Group 3: Golimumab 100 mg | Combined Golimumab
Number analyzed (Participants) | 150 | 147 | 148 | 295
participants | 44 | 82 | 87 | 169
Statistical Analysis 1: Comparison: Group 1: Placebo vs Combined Golimumab; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Stratified by baseline Methorexate (MTX)
Statistical Analysis 2: Comparison: Group 1: Placebo vs Group 2: Golimumab 50 mg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Test was performed because Group 1: Placebo was significantly different from Combined Groups 2 & 3; Stratified by baseline MTX
Statistical Analysis 3: Comparison: Group 1: Placebo vs Group 3: Golimumab 100 mg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Test was performed because Group 1: Placebo was significantly different from Combined Groups 2 & 3; Stratified by baseline MTX

4. Secondary Outcome: American College of Rheumatology (ACR) 20 at Week 24
Description: Number of patients who achieved ACR 20 response at Week (Wk) 24. ACR 20 response is an improvement of >= 20% from baseline in both the tender and swollen joint count and in at least 3 of the 5 assessments ( patient's assessment of pain visual analog scale (VAS), patient's global assessemnt of disease activity VAS scale, Physician's global assessment of disease activity VAS scale,HAQ and CRP)
Time Frame: From Baseline to Week 24
Population: Randomized participants (excluding 1 site). Participants considered non-responders if used any prohibited medications or discontinued SC study agent due to lack of efficacy. Missing ACR components imputed by LOCF unless all components were missing; in which case considered non-responders. Wk 16 ACR response used for change in study tx.
Measure: Number; unit: participants
Arm/Group | Group 1: Placebo | Group 2: Golimumab 50 mg | Group 3: Golimumab 100 mg | Combined Golimumab
Number analyzed (Participants) | 150 | 147 | 148 | 295
participants | 24 | 46 | 63 | 109
Statistical Analysis 1: Comparison: Group 1: Placebo vs Combined Golimumab; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Stratified by baseline Methotrexate (MTX)
Statistical Analysis 2: Comparison: Group 1: Placebo vs Group 2: Golimumab 50 mg; Test type: Superiority or Other; p = 0.002, Cochran-Mantel-Haenszel — Test was performed because Group 1: Placebo was significantly different from Combined Groups 2 & 3; Stratified by baseline MTX
Statistical Analysis 3: Comparison: Group 1: Placebo vs Group 3: Golimumab 100 mg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Test was performed because Group 1: Placebo was significantly different from Combined Groups 2 & 3; Stratified by baseline MTX

5. Secondary Outcome: Health Assessment Questionnaire (HAQ) Score at Week 24
Description: Improvement from baseline in HAQ score at Week 24. This 20-question instrument assesses the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living). Responses in each functional area are scored from 0, indicating no difficulty, to 3, indicating inability to perform a task in that area based on the worst score from the questions that pertain to that task. The HAQ score is determined by the average of the 8 scores; HAQ ranges from 0 to 3.
Time Frame: From Baseline to Week 24
Population: Randomized participants (excluding 1 site). Missing scores imputed by Last Observation Carried Forward. Week 16 scores were used for participants with change in study treatment.
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | Group 1: Placebo | Group 2: Golimumab 50 mg | Group 3: Golimumab 100 mg | Combined Golimumab
Number analyzed (Participants) | 150 | 147 | 148 | 295
scores on a scale | 0.0000 [-0.2500 to 0.2500] | 0.1250 [0.0000 to 0.5000] | 0.2500 [0.0000 to 0.5000] | 0.2500 [0.0000 to 0.5000]
Statistical Analysis 1: Comparison: Group 1: Placebo vs Combined Golimumab; Test type: Superiority or Other; p < 0.001, ANOVA on van der Waerden normal scores; Stratified by baseline Methotrexate (MTX)
Statistical Analysis 2: Comparison: Group 1: Placebo vs Group 2: Golimumab 50 mg; Test type: Superiority or Other; p < 0.001, ANOVA on van der Waerden normal scores. — Test was performed because Group 1: Placebo was significantly different from Combined Groups 2 & 3; Stratified by baseline MTX
Statistical Analysis 3: Comparison: Group 1: Placebo vs Group 3: Golimumab 100 mg; Test type: Superiority or Other; p < 0.001, ANOVA on van der Waerden normal scores. — Test was performed because Group 1: Placebo was significantly different from Combined Groups 2 & 3; Stratified by baseline MTX

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 5 years
Description: Only participants who received at least 1 dose of golimumab were included in the safety analysis. The total number of participants at risk for adverse events is therefore less than the number of participants who started the study.
Groups:
- Group 1: Golimumab 50 mg SC Injections Only: Participants who were treated with golimumab and received golimumab 50 mg injections only during the study.
- Group 2: Golimumab 100 mg SC Injections Only: Participants who were treated with golimumab and received golimumab 100 mg injections only during the study.
- Group 3: Golimumab 50 and 100 mg SC Injections: Participants who were treated with golimumab and received at least one injection of both golimumab 50 mg and golimumab 100 mg during the study.
Arm/Group | Group 1: Golimumab 50 mg SC Injections Only | Group 2: Golimumab 100 mg SC Injections Only | Group 3: Golimumab 50 and 100 mg SC Injections
Serious Adverse Events (participants affected / at risk) | 34/98 | 46/138 | 71/195
Other Adverse Events (participants affected / at risk) | 76/98 | 117/138 | 172/195
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Golimumab 50 mg SC Injections Only (N=98) | Group 2: Golimumab 100 mg SC Injections Only (N=138) | Group 3: Golimumab 50 and 100 mg SC Injections (N=195)
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Acute Coronary Syndrome (Cardiac disorders) | 0 | 0 | 2
Acute Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1
Angina Pectoris (Cardiac disorders) | 0 | 1 | 1
Aortic Valve Incompetence (Cardiac disorders) | 0 | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 1 | 2
Atrial Flutter (Cardiac disorders) | 1 | 0 | 0
Cardiac Failure Congestive (Cardiac disorders) | 0 | 2 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 1
Cardiovascular Disorder (Cardiac disorders) | 0 | 0 | 1
Coronary Artery Disease (Cardiac disorders) | 1 | 0 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 2 | 0
Sick Sinus Syndrome (Cardiac disorders) | 0 | 0 | 1
Supraventricular Tachycardia (Cardiac disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1
Torsade De Pointes (Cardiac disorders) | 0 | 0 | 1
Branchial Cleft Cyst (Congenital, familial and genetic disorders) | 0 | 0 | 1
Adrenal Insufficiency (Endocrine disorders) | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 2
Colitis Ulcerative (Gastrointestinal disorders) | 1 | 0 | 0
Colonic Polyp (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1
Diverticulum Intestinal (Gastrointestinal disorders) | 0 | 0 | 1
Gastric Polyps (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 2
Gastritis Erosive (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal Disorder (Gastrointestinal disorders) | 0 | 0 | 1
Inguinal Hernia (Gastrointestinal disorders) | 0 | 0 | 1
Large Intestine Perforation (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 2 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1 | 1
Splenic Artery Aneurysm (Gastrointestinal disorders) | 0 | 1 | 0
Varices Oesophageal (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0
Chest Pain (General disorders) | 1 | 0 | 0
Device Breakage (General disorders) | 0 | 0 | 1
Device Dislocation (General disorders) | 0 | 1 | 0
Device Failure (General disorders) | 0 | 0 | 1
Generalised Oedema (General disorders) | 0 | 0 | 1
Hernia (General disorders) | 1 | 0 | 0
Multi-Organ Failure (General disorders) | 0 | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 1
Pain (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 1
Bile Duct Stone (Hepatobiliary disorders) | 0 | 0 | 1
Biliary Cirrhosis Primary (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 1
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis Chronic (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 1
Drug-Induced Liver Injury (Hepatobiliary disorders) | 0 | 0 | 1
Abdominal Abscess (Infections and infestations) | 0 | 1 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 2
Cellulitis Streptococcal (Infections and infestations) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 2 | 2
Erysipelas (Infections and infestations) | 0 | 0 | 1
Extradural Abscess (Infections and infestations) | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 2
Gastroenteritis Salmonella (Infections and infestations) | 0 | 1 | 0
Herpes Zoster (Infections and infestations) | 0 | 1 | 0
Histoplasmosis (Infections and infestations) | 0 | 0 | 1
Histoplasmosis Disseminated (Infections and infestations) | 0 | 1 | 0
Infected Skin Ulcer (Infections and infestations) | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 2
Intervertebral Discitis (Infections and infestations) | 1 | 1 | 0
Lung Infection Pseudomonal (Infections and infestations) | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 1
Pelvic Abscess (Infections and infestations) | 0 | 0 | 1
Periorbital Cellulitis (Infections and infestations) | 1 | 1 | 0
Pneumonia (Infections and infestations) | 3 | 5 | 10
Post Procedural Infection (Infections and infestations) | 0 | 0 | 1
Pulmonary Tuberculosis (Infections and infestations) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1 | 0
Salpingitis (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 5
Staphylococcal Abscess (Infections and infestations) | 1 | 1 | 0
Staphylococcal Infection (Infections and infestations) | 0 | 0 | 1
Subcutaneous Abscess (Infections and infestations) | 0 | 1 | 1
Tracheobronchitis (Infections and infestations) | 0 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 2 | 5
Urosepsis (Infections and infestations) | 2 | 0 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1 | 1 | 1
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Fractured Sacrum (Injury, poisoning and procedural complications) | 0 | 1 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 1 | 1
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Meniscus Lesion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Muscle Rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Open Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pelvic Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pubis Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Stress Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound Dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Bone Disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Compartment Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint Effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Mobility Decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 8
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 4 | 2 | 8
Rheumatoid Nodule (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Scleroderma (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Cervix Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Diffuse Large B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung Carcinoma Cell Type Unspecified Stage Iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Squamous Cell Carcinoma of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Thyroid Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Urinary Tract Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Carpal Tunnel Syndrome (Nervous system disorders) | 0 | 0 | 2
Cerebrovascular Accident (Nervous system disorders) | 1 | 3 | 1
Cervicobrachial Syndrome (Nervous system disorders) | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 0 | 1
Demyelination (Nervous system disorders) | 0 | 1 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1
Migraine (Nervous system disorders) | 1 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 0 | 0 | 1
Viith Nerve Paralysis (Nervous system disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1
Mental Status Changes (Psychiatric disorders) | 0 | 1 | 0
Calculus Urinary (Renal and urinary disorders) | 1 | 0 | 0
Renal Disorder (Renal and urinary disorders) | 1 | 0 | 0
Renal Failure (Renal and urinary disorders) | 0 | 0 | 1
Renal Failure Acute (Renal and urinary disorders) | 0 | 1 | 0
Renal Tubular Necrosis (Renal and urinary disorders) | 0 | 0 | 1
Vesical Fistula (Renal and urinary disorders) | 0 | 0 | 1
Endometriosis (Reproductive system and breast disorders) | 0 | 0 | 1
Female Genital Tract Fistula (Reproductive system and breast disorders) | 0 | 0 | 1
Uterine Haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Mediastinal Mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural Fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Drug Detoxification (Surgical and medical procedures) | 1 | 0 | 0
Aortic Thrombosis (Vascular disorders) | 1 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 3 | 0
Haematoma (Vascular disorders) | 0 | 0 | 2
Haemorrhage (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 2
Hypotension (Vascular disorders) | 0 | 1 | 0
Labile Blood Pressure (Vascular disorders) | 1 | 0 | 0
Orthostatic Hypotension (Vascular disorders) | 0 | 0 | 1
Subclavian Artery Stenosis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Golimumab 50 mg SC Injections Only (N=98) | Group 2: Golimumab 100 mg SC Injections Only (N=138) | Group 3: Golimumab 50 and 100 mg SC Injections (N=195)
Vertigo (Ear and labyrinth disorders) | 5 | 4 | 4
Dry Eye (Eye disorders) | 5 | 4 | 5
Diarrhoea (Gastrointestinal disorders) | 4 | 22 | 28
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 6 | 10
Nausea (Gastrointestinal disorders) | 9 | 18 | 21
Vomiting (Gastrointestinal disorders) | 3 | 12 | 7
Fatigue (General disorders) | 2 | 16 | 16
Injection Site Erythema (General disorders) | 6 | 13 | 18
Oedema Peripheral (General disorders) | 3 | 10 | 11
Pyrexia (General disorders) | 2 | 4 | 10
Seasonal Allergy (Immune system disorders) | 2 | 9 | 2
Bronchitis (Infections and infestations) | 11 | 22 | 24
Ear Infection (Infections and infestations) | 2 | 7 | 8
Influenza (Infections and infestations) | 4 | 7 | 15
Nasopharyngitis (Infections and infestations) | 10 | 26 | 37
Oral Herpes (Infections and infestations) | 6 | 9 | 7
Pneumonia (Infections and infestations) | 2 | 7 | 6
Rhinitis (Infections and infestations) | 2 | 9 | 2
Sinusitis (Infections and infestations) | 19 | 23 | 35
Upper Respiratory Tract Infection (Infections and infestations) | 25 | 43 | 49
Urinary Tract Infection (Infections and infestations) | 13 | 12 | 22
Viral Infection (Infections and infestations) | 2 | 7 | 4
Contusion (Injury, poisoning and procedural complications) | 2 | 8 | 12
Excoriation (Injury, poisoning and procedural complications) | 3 | 6 | 10
Laceration (Injury, poisoning and procedural complications) | 2 | 7 | 14
Alanine Aminotransferase Increased (Investigations) | 6 | 0 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 20 | 25
Back Pain (Musculoskeletal and connective tissue disorders) | 8 | 17 | 36
Bursitis (Musculoskeletal and connective tissue disorders) | 4 | 6 | 10
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 | 8 | 3
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 12 | 6
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 | 9 | 15
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 5 | 13
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 4 | 9 | 16
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 14 | 23 | 53
Tendonitis (Musculoskeletal and connective tissue disorders) | 4 | 12 | 16
Dizziness (Nervous system disorders) | 4 | 8 | 10
Headache (Nervous system disorders) | 14 | 14 | 19
Hypoaesthesia (Nervous system disorders) | 2 | 8 | 5
Paraesthesia (Nervous system disorders) | 4 | 8 | 11
Anxiety (Psychiatric disorders) | 1 | 12 | 11
Depression (Psychiatric disorders) | 3 | 8 | 18
Insomnia (Psychiatric disorders) | 0 | 11 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 13 | 24
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 4 | 8 | 15
Rash (Skin and subcutaneous tissue disorders) | 4 | 8 | 19
Hypertension (Vascular disorders) | 10 | 17 | 34

LIMITATIONS AND CAVEATS:
The count of patients with any nonserious adverse events (NAE) excludes patients who only had NAE that occurred in <= 5% of patients. This information may vary from existing approved labeling and publications due to the requirement of this website.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, the only disclosure restriction on the PI is that the sponsor has 60 days to review results communications prior to public release and can embargo communications regarding trial results for a period that does not exceed 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.